CLINICAL TRIAL: NCT00456261
Title: A Randomized Phase II Trial of Pemetrexed/Gemcitabine/Bevacizumab or Pemetrexed/Carboplatin/Bevacizumab in the First-Line Treatment of Elderly Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: First-Line Treatment of A Comparison of 2 Treatments in Elderly Patients With Advanced NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Genentech, Inc. (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI LUN 139
Record Dates: First submitted 2007-04-03; First posted 2007-04-04 (Estimated); Results first posted 2013-02-27 (Estimated); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Lung Cancer
Keywords: Non Small Cell Lung Cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Gemcitabine; Bevacizumab; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort A (Experimental): Cohort A, will receive bevacizumab 10mg/kg by vein over 30-90 minutes followed by pemetrexed 500 mg/m2 by vein over 10 minutes followed by gemcitabine 1500 mg/m2 by vein over 30-60 minutes. This regimen will be given on day 1 and day 15 of each treatment cycle. Each cycle is 28 days long. As long as their disease does not worsen patients can receive up to a maximum of 6 cycles of this combination chemotherapy. Following that they can receive bevacizumab alone once every 2 weeks as long as their disease does not worsen.
  Interventions: Drug: Pemetrexed; Drug: Gemcitabine; Drug: Bevacizumab
- Cohort B (Experimental): Cohort B, will receive bevacizumab 15mg/kg by vein over 30-90 minutes followed by pemetrexed 500 mg/m2 by vein over approximately 10 minutes followed by carboplatin AUC=5 by vein over 30-60 minutes. This regimen will be given on day 1 of each treatment cycle. Each cycle is 21 days long. As long as their disease does not worsen patients can receive up to a maximum of 6 cycles of this combination chemotherapy. Following that they can receive bevacizumab alone once every 3 weeks as long as their disease does not worsen.
  Interventions: Drug: Pemetrexed; Drug: Bevacizumab; Drug: Carboplatin

INTERVENTIONS:
Drug: Pemetrexed — pemetrexed 500 mg/m2
  Other Names: Alimta
Drug: Gemcitabine — gemcitabine 1500 mg/m2
  Other Names: Gemzar
  Arms: Cohort A
Drug: Bevacizumab — bevacizumab 10mg/kg bevacizumab 15mg/kg
  Other Names: Avastin
Drug: Carboplatin — carboplatin AUC=5
  Other Names: Paraplatin
  Arms: Cohort B

SUMMARY:
This trial will look at 2 different drug combinations that have well known safety profiles and are known to be active against non small cell lung cancer and combine them with bevacizumab, an experimental drug that has shown effectiveness when added to other drug combinations for advanced non-small cell lung cancer. The primary objective in this study is to see how well this combination of drugs keeps the cancer from getting worse in this elderly population of non-small cell lung cancer patients.

DETAILED DESCRIPTION:
Patients in this study will be assigned to one of 2 treatment groups. The selection of the treatment groups will be done randomly by a computer.

The first group, Cohort A, will receive bevacizumab 10mg/kg by vein over 30-90 minutes followed by pemetrexed 500 mg/m2 by vein over 10 minutes followed by gemcitabine 1500 mg/m2 by vein over 30-60 minutes. This regimen will be given on day 1 and day 15 of each treatment cycle. Each cycle is 28 days long. As long as their disease does not worsen patients can receive up to a maximum of 6 cycles of this combination chemotherapy. Following that they can receive bevacizumab alone once every 2 weeks as long as their disease does not worsen.

The second group, Cohort B, will receive bevacizumab 15mg/kg by vein over 30-90 minutes followed by pemetrexed 500 mg/m2 by vein over approximately 10 minutes followed by carboplatin AUC=5 by vein over 30-60 minutes. This regimen will be given on day 1 of each treatment cycle. Each cycle is 21 days long. As long as their disease does not worsen patients can receive up to a maximum of 6 cycles of this combination chemotherapy. Following that they can receive bevacizumab alone once every 3 weeks as long as their disease does not worsen.

In both regimens vitamin B12 injections and Folic Acid pills will be given to reduce the occurrence of side effects from the treatment.

Each patient's disease will be evaluated at intervals by the proper scans or X-rays to see how well the cancer is responding to the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-small cell bronchogenic carcinoma, (adenocarcinoma, or large cell carcinoma)
* Patients who have newly diagnosed unresectable stage III or stage IV disease are eligible.
* Must be at least 70 years of age
* Must have measurable disease by CT scan
* Must be able to be up and about and care for themselves
* May not have received prior treatment for stage III or IV disease
* Must have adequate white and red blood cells and platelets.
* Must be able to take Vitamin B12, Folic Acid and dexamethasone as stated in the study
* Must be able to understand the nature of this study and give written informed consent
* Adequate liver and kidney function

Exclusion Criteria:

* Past or current history of cancer with the exception of treated non- melanoma skin cancer or carcinoma in-situ of the cervix, or other cancers cured by local therapy alone and have been disease free for five years
* Female patients who are pregnant or are lactating are ineligible
* History of unstable angina or myocardial infarction within 6 months prior to beginning bevacizumab
* Brain metastasis - cancer that has spread to the brain
* Major surgical procedure, open biopsy, or significant traumatic injury within 6 weeks of beginning bevacizumab or anticipation of need for major surgical procedure during the course of the study
* Full-dose oral or by vein anticoagulation or receiving anti-clotting therapy within 10 days of starting treatment
* Serious nonhealing wound, ulcer, or bone fracture
* Bleeding or clotting disorders
* Uncontrolled high blood pressure or serious heart arrhythmia requiring medication
* History of abdominal fistula, gastrointestinal perforation, or intra- abdominal abscess within 6 months prior to beginning bevacizumab
* Chronic non-steroidal anti-inflammatory use is not allowed on study
* History of stroke or TIAs within the last 6 months

Please Note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 110 (Actual)
Dates: Start 2007-03; Primary Completion 2010-02 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R Spigel, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (18):
- United States (18):
  - Northeast Alabama Regional Medical Center, Anniston, Alabama
  - NEA Baptist Clinic, Jonesboro, Arkansas
  - Florida Cancer Specialists, Fort Myers, Florida
  - Watson Clinic Center for Cancer Care and Research, Lakeland, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Wellstar Cancer Research, Marietta, Georgia
  - Providence Medical Group, Terre Haute, Indiana
  - Graves-Gilbert Clinic, Bowling Green, Kentucky
  - Consultants in Blood Disorders and Cancer, Louisville, Kentucky
  - Mercy Hospital, Portland, Maine
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Methodist Cancer Center, Omaha, Nebraska
  - Cancer Care of Western North Carolina, Asheville, North Carolina
  - Oncology Hematology Care, Cincinnati, Ohio
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Associates in Hematology Oncology, Chattanooga, Tennessee
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee

REFERENCES:
- [Background] Spigel DR, Hainsworth JD, Shipley DL, Ervin TJ, Kohler PC, Lubiner ET, Peyton JD, Waterhouse DM, Burris HA 3rd, Greco FA. A randomized phase II trial of pemetrexed/gemcitabine/bevacizumab or pemetrexed/carboplatin/bevacizumab in the first-line treatment of elderly patients with advanced non-small cell lung cancer. J Thorac Oncol. 2012 Jan;7(1):196-202. doi: 10.1097/JTO.0b013e3182307efe. PMID 21900836

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab/Pemetrexed/Gemcitabine: Cohort A, will receive bevacizumab 10mg/kg by vein over 30-90 minutes followed by pemetrexed 500 mg/m2 by vein over 10 minutes followed by gemcitabine 1500 mg/m2 by vein over 30-60 minutes. This regimen will be given on day 1 and day 15 of each treatment cycle. Each cycle is 28 days long. As long as their disease does not worsen patients can receive up to a maximum of 6 cycles of this combination chemotherapy. Following that they can receive bevacizumab alone once every 2 weeks as long as their disease does not worsen.
- Bevacizumab/Pemetrexed/Carboplatin: Cohort B, will receive bevacizumab 15mg/kg by vein over 30-90 minutes followed by pemetrexed 500 mg/m2 by vein over approximately 10 minutes followed by carboplatin AUC=5 by vein over 30-60 minutes. This regimen will be given on day 1 of each treatment cycle. Each cycle is 21 days long. As long as their disease does not worsen patients can receive up to a maximum of 6 cycles of this combination chemotherapy. Following that they can receive bevacizumab alone once every 3 weeks as long as their disease does not worsen.
Period: Combination Therapy
Arm/Group | Bevacizumab/Pemetrexed/Gemcitabine | Bevacizumab/Pemetrexed/Carboplatin
Started | 55 | 55
Completed | 3 | 29
Not Completed | 52 | 26
Period: Maintenance Therapy
Arm/Group | Bevacizumab/Pemetrexed/Gemcitabine | Bevacizumab/Pemetrexed/Carboplatin
Started | 3 | 29
Completed | 3 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bevacizumab/Pemetrexed/Gemcitabine | Bevacizumab/Pemetrexed/Carboplatin | Total
Number analyzed (Participants) | 55 | 55 | 110
Age, Continuous [Median (Full Range); unit: years] | 76 [70 to 89] | 77 [70 to 88] | 77 [70 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 29 | 55
  Male | 29 | 26 | 55
Region of Enrollment [Number; unit: participants]
  United States | 55 | 55 | 110

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression (TTP), the Length of Time, in Months, That Patients Were Alive From Their First Date of Protocol Treatment Until Worsening of Their Disease
Description: Time to Progression (TTP) is defined as the interval between the date of treatment initiation and the date of progressive disease. Progression is defined using the Response Evaluation Criteria in Solid Tumors (RECIST v1.0). Progressive Disease (PD): At least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or unequivocal progression of non-target lesions or the appearance of one or more new lesions.
Time Frame: From the date of treatment initiation until the date of first documented PD or date of last study contact or date of other therapy begins up to 18 months
Population: All patients were analyzed for a response by RECIST v1.0. Intent to treat efficacy analysis set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab/Pemetrexed/Gemcitabine | Bevacizumab/Pemetrexed/Carboplatin
Number analyzed (Participants) | 55 | 55
months | 4.7 [3.8 to 5.8] | 10.2 [6.3 to 12.7]

2. Secondary Outcome: Overall Response Rate (ORR), the Percentage of Patients Who Experience an Objective Benefit From Treatment
Description: Overall response rate (ORR) is defined as the percentage of patients who have a partial or complete response to therapy. Responses were assessed by the Response Evaluation Criteria in Solid Tumors (RECIST; version 1.0). Complete Response: Disappearance of all target lesions, and disappearance of all non-target lesions. Partial Response: At least a 30% decrease in the sum of the longest diameter of target lesions (taking as reference the baseline sum of longest diameters)
Time Frame: From date of treatment initiation to end of study treatment up to 18 months
Population: All patients were analyzed for a response by RECIST v1.0. Intent to treat analysis set.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Bevacizumab/Pemetrexed/Gemcitabine | Bevacizumab/Pemetrexed/Carboplatin
Number analyzed (Participants) | 55 | 55
percentage of patients | 35 [23 to 49] | 35 [23 to 49]

3. Secondary Outcome: Overall Survival (OS), the Length of Time, in Months, That Patients Were Alive From Their First Date of Protocol Treatment Until Death
Description: OS is defined as the time from the date of study entry until the date of death due to any cause. In the absence of confirmation of death or lack of data beyond follow-up period, the survival time was censored to the last date the participant was known to be alive.
Time Frame: From date of study entry until the date of death from any cause or the date the patient was last known alive, up to 18 months
Population: All patients were included in the analysis. Intent to treat analysis set.
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab/Pemetrexed/Gemcitabine | Bevacizumab/Pemetrexed/Carboplatin
Number analyzed (Participants) | 55 | 55
months | 7.5 [5.6 to 11.3] | 14.8 [10.25 to NA] — Upper limit not reached due to patients continuing treatment at time of analysis.

ADVERSE EVENTS:
Arm/Group | Bevacizumab/Pemetrexed/Gemcitabine | Bevacizumab/Pemetrexed/Carboplatin
Serious Adverse Events (participants affected / at risk) | 33/55 | 21/55
Other Adverse Events (participants affected / at risk) | 55/55 | 55/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab/Pemetrexed/Gemcitabine (N=55) | Bevacizumab/Pemetrexed/Carboplatin (N=55)
Hemorrhage - Pulmonary (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Thrombosis/Thrombus/Embolism (Vascular disorders) | 3 (3) | 1 (1)
Infection - Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death - disease progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Pulmonary - COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (4)
Perforation - Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Febrile neutropenia (Infections and infestations) | 2 (2) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Neutrophils (Immune system disorders) | 3 (3) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Infection - Pneumonia (Infections and infestations) | 7 (8) | 1 (1)
Multi-system Organ Failure (General disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 1 (1) | 1 (1)
Hypertension (Cardiac disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0)
CNS Cerebrovascular ischemia (Nervous system disorders) | 2 (2) | 1 (1)
Cardiopulmonary Arrest (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular Arrhythmia - Ventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Infection - gangrene (Infections and infestations) | 1 (1) | 0 (0)
Infection - cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Platelets (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
ARDS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Perforation - duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Confusion (Nervous system disorders) | 1 (1) | 0 (0)
Supraventricular arrhythmia - Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Infection with Normal ANC (Infections and infestations) | 1 (1) | 0 (0)
Pain - rectum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain - Abdomen (General disorders) | 1 (1) | 0 (0)
GI Other - strangulated inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pericardial Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1) | 2 (2)
Obstruction, GU - Bladder (Renal and urinary disorders) | 0 (0) | 1 (1)
Cardiac Ischemia/Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Pain - joint (General disorders) | 0 (0) | 1 (1)
Dysphagia (General disorders) | 0 (0) | 1 (1)
Aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Infection - methicillin-resistant staphylococcus aureas (Infections and infestations) | 0 (0) | 1 (1)
Infection - urinary tract (Infections and infestations) | 1 (1) | 0 (0)
Ulcer - stomach (Gastrointestinal disorders) | 1 (1) | 0 (0)
Consitutional symptoms, other - failure to thrive (General disorders) | 1 (1) | 0 (0)
Disease progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytes (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab/Pemetrexed/Gemcitabine (N=55) | Bevacizumab/Pemetrexed/Carboplatin (N=55)
Alkaline Phosphatase (Metabolism and nutrition disorders) | 9 (13) | 6 (11)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (5) | 6 (17)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 9 (34)
ALT (Metabolism and nutrition disorders) | 10 (17) | 5 (7)
Anorexia (Gastrointestinal disorders) | 25 (55) | 26 (65)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (12) | 14 (33)
AST (Metabolism and nutrition disorders) | 13 (27) | 7 (7)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 7 (12)
Confusion (Nervous system disorders) | 5 (7) | 0 (0)
Constipation (Gastrointestinal disorders) | 21 (34) | 22 (77)
Cough (Respiratory, thoracic and mediastinal disorders) | 21 (36) | 20 (68)
Creatinine (Metabolism and nutrition disorders) | 3 (5) | 8 (11)
Dehydration (Gastrointestinal disorders) | 14 (18) | 8 (16)
Dermatology - Other (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4) — Laceration
Diarrhea (Gastrointestinal disorders) | 14 (22) | 19 (40)
Dizziness (Nervous system disorders) | 11 (16) | 16 (22)
Dry Eye (Eye disorders) | 3 (4) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 4 (6) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 4 (9)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 34 (69) | 29 (109)
Edema - Limb (Blood and lymphatic system disorders) | 16 (33) | 10 (26)
Erythema (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (7)
Fatigue (General disorders) | 46 (158) | 48 (298)
Fever (General disorders) | 16 (17) | 3 (3)
Febrile Neutropenia (Infections and infestations) | 4 (4) | 0 (0)
Pain - Head (General disorders) | 8 (10) | 14 (41)
Neutrophils (Blood and lymphatic system disorders) | 39 (84) | 42 (118)
Hemoglobin (Blood and lymphatic system disorders) | 45 (128) | 45 (243)
Platelets (Blood and lymphatic system disorders) | 30 (55) | 40 (153)
Leukocytes (Blood and lymphatic system disorders) | 39 (89) | 47 (151)
Respiratary - Other (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 0 (0) — Hemoptysis
Hemorrhage - Nose (Blood and lymphatic system disorders) | 10 (21) | 15 (26)
Voice Changes (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (8)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 4 (6)
Hyperglycemia (Metabolism and nutrition disorders) | 15 (28) | 15 (32)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 6 (18)
Hypertension (Cardiac disorders) | 7 (13) | 18 (42)
Hypoalbuminemia (Metabolism and nutrition disorders) | 11 (19) | 9 (21)
Hypocalcemia (Metabolism and nutrition disorders) | 7 (9) | 4 (7)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 15 (32)
Hypokalemia (Metabolism and nutrition disorders) | 3 (4) | 6 (14)
Hyponatremia (Metabolism and nutrition disorders) | 7 (18) | 10 (14)
Hypotension (Cardiac disorders) | 3 (3) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 0 (0)
Infection - NOS (Infections and infestations) | 30 (61) | 17 (31)
Insomnia (General disorders) | 10 (19) | 7 (12)
INR (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Mood Alteration - Anxiety (Psychiatric disorders) | 4 (4) | 3 (7)
Mood Alteration - Depression (Psychiatric disorders) | 3 (5) | 4 (14)
Mucositis/Stomatitis (Gastrointestinal disorders) | 6 (8) | 11 (20)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 18 (35)
Nasal/Paranasal Reactions (Respiratory, thoracic and mediastinal disorders) | 9 (20) | 3 (9)
Nausea (Gastrointestinal disorders) | 29 (46) | 29 (66)
Neuropathy - Sensory (Nervous system disorders) | 5 (10) | 4 (5)
Pain - NOS (General disorders) | 0 (0) | 4 (14)
Pain - Abdomen (General disorders) | 7 (17) | 4 (5)
Pain - Back (General disorders) | 0 (0) | 4 (6)
Pain - Bone (General disorders) | 0 (0) | 3 (5)
Pain - Chest (General disorders) | 4 (5) | 11 (23)
Pain - Limb (General disorders) | 4 (4) | 6 (12)
Pain - Mouth (General disorders) | 3 (9) | 3 (9)
Pain - Neck (General disorders) | 0 (0) | 3 (9)
Proteinuria (Renal and urinary disorders) | 22 (42) | 28 (119)
Pruritis (Skin and subcutaneous tissue disorders) | 4 (4) | 5 (6)
Pulmonary - COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 0 (0)
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 15 (25) | 16 (32)
ARDS (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Rigor/Chills (General disorders) | 7 (13) | 0 (0)
Taste Alteration (Gastrointestinal disorders) | 5 (8) | 12 (40)
Thrombosis/Thrombus/Embolism (Vascular disorders) | 6 (10) | 4 (5)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 3 (6)
Voice Changes (General disorders) | 0 (0) | 9 (36)
Vomiting (Gastrointestinal disorders) | 6 (7) | 13 (18)
Watery Eye (Eye disorders) | 0 (0) | 5 (15)
Weight Loss (Metabolism and nutrition disorders) | 9 (15) | 9 (29)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites